CLINICAL TRIAL: NCT05140876
Title: Supporting Treatment Adherence for Resilience and Thriving
Brief Title: Supporting Treatment Adherence for Resilience and Thriving (START)
Acronym: START
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor and Chair, Florida International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20190578; R01DA049843 (NIH)
Record Dates: First submitted 2021-11-15; First posted 2021-12-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Adherence, Medication; HIV-1-infection; Stimulant Use
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START mHealth Intervention (Experimental): Participants randomized to receive the START mHealth intervention will have access to the mHealth application for 6 months following randomization.
  Interventions: Behavioral: START mHealth Intervention
- Website referrals (No Intervention): Participants in this condition will receive no intervention and will have access to a website with resources related to substance use disorder treatment and HIV treatment.

INTERVENTIONS:
Behavioral: START mHealth Intervention — The START mHealth intervention is a mobile application that will be downloaded by participants through their mobile phones. The application targets information, motivation, and behavioral skills relevant to ART adherence. Participants will have access to this application for 6 months.
  Arms: START mHealth Intervention

SUMMARY:
This Phase II randomized controlled trial is testing the efficacy of a cell phone application called START for helping men who use stimulants like methamphetamine to get the most out of their HIV treatment.

ELIGIBILITY:
1. Assigned male at birth;
2. Identifies as male;
3. Age 18 or older;
4. Reads and speaks English;
5. Continental US residency;
6. Reports ever having had anal sex with a man;
7. Self-reported HIV diagnosis for 3 or more months and currently taking anti-retroviral therapy (ART)
8. Reports a detectable viral load during past year OR no viral load test in the past 10+ months OR reports < 90% adherence to ART;
9. Screens positive for a moderate or severe stimulant use disorder in the past 3 months with an abbreviated version of the National Institute on Drug Abuse (NIDA)-modified Alcohol, Smoking and Substance. Involvement Screening Test (ASSIST);
10. Has an iPhone or Android smartphone;
11. Is willing to participate in an mHealth intervention

Exclusion Criteria:

1. HIV-negative or never tested for HIV;
2. HIV-positive men without a current ART prescription;
3. Does not return a viable DBS specimen at baseline for viral load testing
4. Not a sexual minority man

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as male
Enrollment: 286 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Unsuppressed HIV Viral Load | 6 Months
  Proportion of participants with a viral load > 300 copies/mL from dried blood spot samples

SECONDARY OUTCOMES:
Unsuppressed Viral Load | 12 Months
  Proportion of participants with a viral load > 300 copies/mL from dried blood spot samples
Self-Reported Stimulant Use Severity | 12 Months
  The Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) provides validated composite scores indexing the severity of cocaine and amphetamine use (Mild = 0-3; Moderate = 4-26; Severe = 27 or greater).
Self-Reported Anti-Retroviral Therapy (ART) Adherence | 12 Months
  Participants will rate on a visual analogue scale the percentage (0% meaning no adherence to 100% meaning complete adherence) of ART medications that they took in the past 30 days
Positive Affect | 12 Months
  Mean positive affect score as measured by the modified Differential Emotions Scale (Range 0-104) with higher scores being indicative of higher positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, PhD, Principal Investigator — Florida International University
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis-Ewart L, Atkins L, Ghanooni D, Diaz JE, Chuku CC, Balise R, DeVries BA, Miller-Perusse M, Ackley Iii D, Moskowitz JT, McCollister K, Fardone E, Hirshfield S, Horvath KJ, Carrico AW. Supporting treatment adherence for resilience and thriving (START): protocol for a mHealth randomized controlled trial. BMC Public Health. 2024 Aug 29;24(1):2350. doi: 10.1186/s12889-024-19745-7. PMID 39210314